CLINICAL TRIAL: NCT04119102
Title: Open Label Study Evaluating DUOBRII in Psoriasis Patients Being Treated With Biologic Agents.
Brief Title: Duobrii in Combination With Biologics
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Psoriasis Treatment Center of Central New Jersey (Other)
Collaborators: Ortho Dermatologics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTC07
Record Dates: First submitted 2019-10-03; First posted 2019-10-08 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Intervention Model Description: open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Open Label Duobrii (Experimental): Duobrii QD
  Interventions: Drug: Duobrii

INTERVENTIONS:
Drug: Duobrii — duobrii applied daily for 4 weeks followed by every other day for 4 weeks.

SUMMARY:
12 weeks DUOBRII to patients with 2%-10% BSA who are receiving biologic therapy for at least 24 weeks

DETAILED DESCRIPTION:
A single center, pilot study of 25 subjects to assess 12 weeks DUOBRII to patients with 2%-10% body surface area who are receiving biologic therapy for at least 24 weeks

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adult ≥ 18 years of age;
2. Diagnosis of chronic plaque-type
3. Psoriasis affecting 2%-10% BSA
4. Patient is being treated with biologic therapy for a minimum of 24 weeks
5. Able and willing to give written informed consent prior to performance of any study-related procedures

Exclusion Criteria:

1. Psoriasis affecting ˂2% or >10% BSA
2. Patient not receiving a biologic agent, or receiving biologic agent <24weeks
3. Received treatment with any topical antipsoriatic drug product within 14 days prior to the Baseline visit.
4. Has previously used DUOBRII

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2019-10-14 (Actual); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Body surface area improvement | 8 weeks
  body surface area determined by palm method where 1 palm is equivalent to 1%

CONTACTS AND LOCATIONS:
Locations (1):
- Psoriasis Treatment Center of Central New Jersey, East Windsor, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No